CLINICAL TRIAL: NCT04128176
Title: An Open-Label Study to Evaluate the Efficacy and Safety of Rituximab Combined With Omalizumab in Patients With Bullous Pemphigoid
Brief Title: Efficacy and Safety of Rituximab Combined With Omalizumab in Patients With Bullous Pemphigoid
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI did not pursue this study; this study was not IRB-approved and never started.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1510820
Record Dates: First submitted 2019-10-12; First posted 2019-10-16 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Bullous Pemphigoid
Keywords: Omalizumab; Rituximab; Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rituximab combined with Omalizumab (Experimental): All patients will receive daily doxycycline, nicotinamide, and high-potency topical steroids. Additionally, all patients will receive rituximab combined with omalizumab.
  Interventions: Drug: Rituximab combined with Omalizumab

INTERVENTIONS:
Drug: Rituximab combined with Omalizumab — Rituximab 1000 mg will be administered by IV infusion 6 months after the patient's initial cycle of rituximab (received in the screening period).Omalizumab (300 mg) will be administered subcutaneously every 2 weeks starting on Day 1 until week 24 (primary endpoint) and again until week 52 (secondary endpoint).
  Other Names: Xolair

SUMMARY:
To evaluate the efficacy of rituximab combined with omalizumab in achieving sustained complete remission, evaluated by Bullous Pemphigoid Disease Area Index (BPDAI) in patients with bullous pemphigoid (BP) at Week 24 in patients with active moderate-to-severe BP refractory to rituximab therapy alone.

DETAILED DESCRIPTION:
This is an open-label, noncontrolled, single center prospective study to evaluate the efficacy and safety of rituximab combined with omalizumab in patients with active moderate-to-severe BP refractory to rituximab treatment alone. Patients must have a confirmed diagnosis of BP and evidence of refractory disease after initiation of rituximab treatment at least 8 weeks prior.

Refractory disease will be defined as a failure of therapy (development of new non-transient lesions or continued extension of old lesions, or failure of established lesions to begin to heal or continued pruritus) or evidence of a relapse/flare (Appearance of ≥3 new lesions/month (blisters, eczematous lesions, or urticarial plaques) or at least one large (>10 cm diameter) eczematous lesion or urticarial plaques that do not heal within 1 week, or extension of established lesions or daily pruritus in patient who have achieved disease control) based on the outcome measures defined for BP from an international panel of experts.41

This study will be conducted at the University of California, Davis Department of Dermatology's investigational site.

The study will consist of 3 periods: a screening period, 24-week treatment period, and a 28-week follow-up period. During the treatment period, patient visits will be monthly. After the primary endpoint at Week 24, follow up assessments will be scheduled every 3 months.

Rituximab 1000 mg will be administered by IV infusion 6 months after the patient's initial cycle of rituximab (received in the screening period). In order to reduce the frequency and severity of infusion-related reactions, all patients will be pre-medicated per the infusion center's therapy beacon protocol. Omalizumab (300 mg) will be administered subcutaneously every 2 weeks starting on Day 1.

All patients will be provided topical clobetasol 0.05% ointment or equivalent strength potency topical corticosteroid. Topical steroid application will be used 40 grams twice daily as needed for itch.

Patients can be discontinued from study treatment at any time during the study. Patients who withdraw from the treatment period will return to the clinic for an early withdrawal visit. After the withdrawal visit, the patient will be asked to enter the follow up period of the study.

From Week 1 through Week 52, patients who do not experience 50% improvement in their BPDAI at week 16 are eligible to receive rescue therapy with prednisone, another immunosuppressive medication (e.g. cellcept), IV Ig, or another treatment or procedure as per the investigator's best medical judgment. Patients who receive rescue therapy will be withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18-90 years of age
* All individuals must have the ability to provide inform consent
* Patients diagnosed with bullous pemphigoid by biopsy, serum ELISA, direct immunofluorescence, indirect immunofluorescence
* Presence of moderate-to-severe active disease refractory to at least one cycle of rituximab therapy

Exclusion Criteria:

* Diagnosis of mucous membrane pemphigoid or evidence of other non-BP autoimmune blistering disease
* Individuals with allergic reaction or adverse reaction to humanized or murine monoclonal antibodies, or known hypersensitivity to any component of rituximab or omalizumab
* Evidence of acute infection or history of a chronic infection including viral hepatitis, recurrent HSV, AIDS, etc
* Women who are pregnant or actively nursing
* Evidence of any new or uncontrolled concomitant disease that, in the investigator's judgment, would preclude patient participation, including but not limited to cardiovascular, pulmonary, nervous system, renal, hepatic, endocrine, malignant, or gastrointestinal disorders
* Treatment with a live or attenuated vaccine within 28 days prior to first rituximab infusion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03 (Estimated); Primary Completion 2023-05-25 (Estimated); Study Completion 2023-11-25 (Estimated)

PRIMARY OUTCOMES:
Disease Remission | 24 weeks
  Complete remission is defined as achieving wound healing with no new active lesions (i.e. Bullous Pemphigoid Disease Area Index (BPDAI) score of 0) for at least 2 consecutive weeks during the 24-week treatment period. BPDAI scores can range from 0 to 360, with lower scores indicating less disease activity and better outcomes.

SECONDARY OUTCOMES:
Disease Remission | 52 weeks
  Proportion of patients achieving a sustained complete remission with rituximab combined with omalizumab at week 52
Number of Disease Flares | 52 weeks
  Total number of disease flares during the treatment period, as defined by appearance of three or more new lesions a month or at least one large (>10 cm diameter) eczematous lesion or urticarial plaques that do not heal within 1 week or by the extension of established lesions.
Time to Remission | 52 weeks
  Time to sustained complete remission
Time to Flares | 52 weeks
  Time to disease flare
Duration of Remission | 52 weeks
  Duration of sustained complete remission
Clinical Impression | 52 weeks
  Clinician impression of change in patients' BP symptoms, as measured by the Clinician Global Impression of Change (CGIC) score during the treatment period. The CGIC is a seven point scale to rate the severity of a patient's illness at the time of the assessment, with higher scores indicating better outcomes.
Patient Impression | 52 weeks
  Patients' impression of change in BP symptoms, as measured by the Patient Global Impression of Change (PGIC) score during the treatment period. The CGIC is a seven point scale to rate the severity of a patient's illness at the time of the assessment, with higher scores indicating better outcomes.
Improvement in Itch | 52 weeks
  Change in patients' scores in improvement of Itch Numeric Rating Scale (NRS) during the treatment period. The NRS is on a scale of 0 to 10 with 0 representing "no itch" and better outcomes.
Health-Related Quality of Life | 52 weeks
  Change in health-related quality of life, as measured by the Dermatology Life Quality Index (DLQI) score from baseline to Week 24. The DLQI is a ten item questionnaire with a sum total of 30 points. The higher the score, the more quality of life is impaired, indicating worse outcomes.

OTHER OUTCOMES:
Adverse Events That Are Related to Treatment | 52 weeks
  To evaluate the safety of rituximab combined with omalizumab by monitoring adverse events related to treatment, such as number of abnormal laboratory values.
Gene Expression | 52 weeks
  To evaluate gene expression profiling of skin biopsies taken (1) before omalizumab therapy and (2) after omalizumab therapy.
Cumulative Corticosteroid Application | 52 weeks
  To evaluate total cumulative dose of topical corticosteroid applied during treatment and follow up periods

CONTACTS AND LOCATIONS:
Overall Officials: Emanual Maverakis, MD, Principal Investigator — UC Davis
Locations (1):
- University of California, Davis, Department of Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ujiie H, Nishie W, Shimizu H. Pathogenesis of bullous pemphigoid. Dermatol Clin. 2011 Jul;29(3):439-46, ix. doi: 10.1016/j.det.2011.03.008. PMID 21605809
- [Background] Maglie R, Hertl M. Pharmacological advances in pemphigoid. Curr Opin Pharmacol. 2019 Jun;46:34-43. doi: 10.1016/j.coph.2018.12.007. Epub 2019 Feb 13. PMID 30769277